CLINICAL TRIAL: NCT07174544
Title: Mobile Self-Management Program Integrating Positive Psychology and Behavioral Activation for Stress Reduction in Young Adults: A Community-Based Randomized Controlled Trial
Brief Title: Mobile Self-Management Program for Stress Reduction in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Hyunjoo Na, Associate professor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MC23FNSI0059; NRF-2022R1A2C1011568 (Other Grant/Funding Number: National Research Foundation of Korea)
Record Dates: First submitted 2025-09-11; First posted 2025-09-16 (Actual); Results first posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Stress (Psychology)
Keywords: Stress; Resilience; Self-Management; Positive Psychology; Mobile Applications; Young Adult
MeSH Terms: interventions — Psychology, Positive

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants receive a mobile self-management intervention that integrates Positive Psychology and Behavioral Activation. The program includes 4 weeks of guided sessions followed by 4 weeks of self-directed use.
  Interventions: Behavioral: Mobile Self-Management Program integrated with Positive Psychology and Behavioral Activation
- Wait-list Control (No Intervention): Participants do not receive the intervention during the first 8 weeks but are offered access to the program after the study period.

INTERVENTIONS:
Behavioral: Mobile Self-Management Program integrated with Positive Psychology and Behavioral Activation — The mobile self-management program consisted of a 4-week guided intervention phase followed by a 4-week self-directed period to encourage continued use. The guided phase was organized around weekly objectives: (1) experiencing positive affect, (2) identifying personal strengths, (3) applying strengths in daily life, and (4) planning a positive future. Program activities included emotional check-ins, gratitude journaling, mindfulness practice, positive behavioral tasks, and goal setting. During the self-directed phase (Weeks 5-8), participants selected from 10 recommended activities tailored to their strengths, promoting sustained engagement and self-management. The program integrated Positive Psychology and Behavioral Activation strategies to reduce stress, enhance resilience, and foster positive behavioral change.
  Arms: Intervention group

SUMMARY:
The goal of this clinical trial is to learn if a mobile self-management program that combines Positive Psychology (PP) and Behavioral Activation (BA) helps reduce stress in young adults in South Korea. It will also examine how the program affects depression, anxiety, and resilience.

The main questions it aims to answer are:

Does the program lower stress levels in young adults with high stress?

Does the program improve other aspects of mental health, such as depression, anxiety, and resilience?

Researchers will compare the mobile program to a wait-list control group to see if the program works to improve stress management.

Participants will:

Be randomly assigned to either the program group or a wait-list control group

Use the mobile program for 4 weeks with guided activities, followed by 4 weeks of self-directed use

Complete surveys at the start, week 2, week 4, and week 8 about their stress, depression, anxiety, and resilience

ELIGIBILITY:
Inclusion Criteria:

* Age 19-34 years at the time of participation
* Proficiency in using digital devices
* Use of an Android-based smartphone or tablet
* Score of ≥14 on the Perceived Stress Scale-10 (PSS-10)
* Provision of informed consent for random assignment

Exclusion Criteria:

* Score <14 on the Perceived Stress Scale-10 (PSS-10)
* Declines random assignment

Ages: 19 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 211 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-08-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- College of Nursing, The Catholic University of Korea, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
The study's informed consent form restricts use of data to this research only. Therefore, IPD will not be shared with other researchers.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: a score of ≥14 on the Perceived Stress Scale-10 (PSS-10)
Period: Overall Study
Arm/Group | Intervention Group | Wait-list Control
Started | 92 | 87
2week | 68 | 80
4week | 53 | 75
8week | 49 | 72
Completed | 49 | 72
Not Completed | 43 | 15
Not completed — Lost to Follow-up | 43 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Wait-list Control | Total
Number analyzed (Participants) | 92 | 87 | 179
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 92 | 87 | 179
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.85 (4.16) | 27.46 (4.42) | 27.66 (4.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 72 | 151
  Male | 13 | 15 | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 92 | 87 | 179
Stress [Mean (Standard Deviation); unit: units on a scale] | 22.64 (5.82) | 19.76 (3.64) | 21.24 (5.08)

OUTCOME MEASURES:

1. Secondary Outcome: Stress at Baseline
Description: Stress was measured using the Korean version of the Perceived Stress Scale - 10 items (PSS-10). The total score ranges from 0 to 40, with higher scores indicating greater perceived stress. Although the scale does not provide a standardized cut-off, prior studies have used a score of 14 or higher to define moderate-to-high levels of stress, and this threshold was applied in the present study.
Time Frame: Baseline
Population: Participants with available PSS-10 data at baseline were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Wait-list Control
Number analyzed (Participants) | 92 | 87
score on a scale | 22.64 (5.82) | 19.76 (3.64)

2. Secondary Outcome: Stress at Week 2
Description: as for outcome 1
Time Frame: Week 2
Population: Participants with available PSS-10 data at week 2 were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Wait-list Control
Number analyzed (Participants) | 68 | 80
score on a scale | 20.57 (5.78) | 19.00 (3.98)

3. Secondary Outcome: Stress at Week 4
Description: as for outcome 1
Time Frame: Week 4
Population: Participants with available PSS-10 data at week 4 were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Wait-list Control
Number analyzed (Participants) | 53 | 75
score on a scale | 20.08 (6.62) | 18.71 (4.00)

4. Secondary Outcome: Depression (PHQ-9) at Baseline
Description: Depression was assessed using the Korean version of the Patient Health Questionnaire-9 items (PHQ-9). The PHQ-9 consists of nine items rated on a 4-point Likert scale (0 = not at all to 3 = nearly every day), assessing symptom frequency over the past two weeks. The total score ranges from 0 to 27, with higher scores indicating more severe depression.
Time Frame: Baseline
Population: Participants with available PHQ-9 data at baseline were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Wait-list Control
Number analyzed (Participants) | 92 | 87
score on a scale | 10.21 (5.89) | 9.24 (5.42)

5. Secondary Outcome: Depression (PHQ-9) at Week 2
Description: as for outcome 4
Time Frame: Week 2
Population: Participants with available PHQ-9 data at week 2 were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Wait-list Control
Number analyzed (Participants) | 68 | 80
score on a scale | 8.34 (5.44) | 8.51 (5.63)

6. Secondary Outcome: Depression (PHQ-9) at Week 4
Description: as for outcome 4
Time Frame: Week 4
Population: Participants with available PHQ-9 data at week 4 were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Wait-list Control
Number analyzed (Participants) | 53 | 75
score on a scale | 7.72 (5.91) | 7.95 (5.36)

7. Primary Outcome: Stress at Week 8
Description: as for outcome 1
Time Frame: Week 8
Population: Participants with available PSS-10 data at week 8 were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Wait-list Control
Number analyzed (Participants) | 49 | 72
score on a scale | 19.41 (6.20) | 18.35 (4.05)
Statistical Analysis 1: Comparison: Intervention Group vs Wait-list Control; Test type: Superiority — Superiority was assessed by comparing outcomes between the intervention and wait-list control groups over time; Generalized estimating equations (GEE); Generalized estimating equations were used to examine changes in outcomes over time between groups, accounting for repeated measurements; Analyses followed the intention-to-treat principle using available data at each assessment time point. Descriptive statistics were used to summarize baseline characteristics

8. Secondary Outcome: Depression (PHQ-9) at Week 8
Description: as for outcome 4
Time Frame: Week 8
Population: Participants with available PHQ-9 data at week 8 were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Wait-list Control
Number analyzed (Participants) | 49 | 72
score on a scale | 8.37 (6.38) | 7.69 (5.50)

9. Secondary Outcome: Anxiety (GAD-7) at Baseline
Description: Anxiety was measured using the Korean version of the Generalized Anxiety Disorder-7 items (GAD-7). The GAD-7 consists of seven items rated on a 4-point Likert scale (0 = not at all to 3 = nearly every day), assessing symptom frequency over the past two weeks. The total score ranges from 0 to 21, with higher scores indicating more severe anxiety.
Time Frame: Baseline
Population: Participants with available GAD-7 data at baseline were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Wait-list Control
Number analyzed (Participants) | 92 | 87
score on a scale | 8.20 (5.75) | 7.68 (4.88)

10. Secondary Outcome: Anxiety (GAD-7) at Week 2
Description: as for outcome 9
Time Frame: Week 2
Population: Participants with available GAD-7 data at week 2 were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Wait-list Control
Number analyzed (Participants) | 68 | 80
score on a scale | 6.88 (5.65) | 7.13 (5.23)

11. Secondary Outcome: Anxiety (GAD-7) at Week 4
Description: as for outcome 9
Time Frame: Week 4
Population: Participants with available GAD-7 data at week 4 were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Wait-list Control
Number analyzed (Participants) | 53 | 75
score on a scale | 6.43 (5.61) | 7.03 (5.21)

12. Secondary Outcome: Anxiety (GAD-7) at Week 8
Description: as for outcome 9
Time Frame: Week 8
Population: Participants with available GAD-7 data at week 8 were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Wait-list Control
Number analyzed (Participants) | 49 | 72
score on a scale | 7.63 (6.11) | 6.36 (4.87)

13. Secondary Outcome: Resilience ( BRS) at Baseline
Description: Resilience was assessed using the Korean version of the Brief Resilience Scale (BRS). The BRS consists of six items rated on a 5-point Likert scale (1 = strongly disagree to 5 = strongly agree). Total scores range from 6 to 30, with higher scores indicating greater resilience.
Time Frame: Baseline
Population: Participants with available BRS data at baseline were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Wait-list Control
Number analyzed (Participants) | 92 | 87
score on a scale | 15.24 (5.06) | 17.79 (1.71)

14. Secondary Outcome: Resilience (BRS) at Week 2
Description: as for outcome 13
Time Frame: Week 2
Population: Participants with available BRS data at week 2 were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Wait-list Control
Number analyzed (Participants) | 68 | 80
score on a scale | 15.37 (5.10) | 17.59 (1.76)

15. Secondary Outcome: Resilience (BRS) at Week 4
Description: as for outcome 13
Time Frame: Week 4
Population: Participants with available BRS data at week 4 were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Wait-list Control
Number analyzed (Participants) | 53 | 75
score on a scale | 16.06 (5.68) | 17.87 (1.93)

16. Secondary Outcome: Resilience (BRS) at Week 8
Description: as for outcome 13
Time Frame: Week 8
Population: Participants with available BRS data at week 8 were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Wait-list Control
Number analyzed (Participants) | 49 | 72
score on a scale | 16.14 (5.87) | 17.54 (1.85)

ADVERSE EVENTS:
Time Frame: From enrollment until completion of the 8-week study period.
Description: All-cause mortality, serious adverse events, and other (non-serious) adverse events were monitored through non-systematic self-report during the study period. This was a non-clinical, community-based behavioral intervention delivered via a mobile self-management program without medical procedures or pharmacological treatment. Therefore, No adverse events were reported in either group.
Arm/Group | Intervention Group | Wait-list Control
All-Cause Mortality (participants affected / at risk) | 0/92 | 0/87
Serious Adverse Events (participants affected / at risk) | 0/92 | 0/87
Other Adverse Events (participants affected / at risk) | 0/92 | 0/87

LIMITATIONS AND CAVEATS:
A key limitation of this study was participant attrition during the 8-week intervention period, as some participants did not complete all weekly or follow-up surveys. This loss to follow-up may have limited the ability to fully determine the intervention's effect over time and reduced the precision of longitudinal comparisons between groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-30): https://cdn.clinicaltrials.gov/large-docs/44/NCT07174544/Prot_SAP_000.pdf